CLINICAL TRIAL: NCT03554837
Title: A Multicenter, Prospective, Non-interventional, Cohort Study to Evaluate the Safety and Effectiveness of Low Dose Edoxaban in Patients With Non-valvular Atrial Fibrillation (NVAF), Who Are Applicable to Any of the Dose Reduction Criteria
Brief Title: Safety and Effectiveness of Low Dose Edoxaban in Patients With NVAF
Acronym: LEDIOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Keun On, Professor, Samsung Medical Center
Other Study IDs: IRB 2017-12-051
Record Dates: First submitted 2018-04-19; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation
Keywords: safety; effectiveness; low dose
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The efficacy and safety of edoxaban has not been adequately studied in Asians versus non-Asians, who are quite different physiologically from each other. Compared with non-East Asian patients, the East Asia patients were twice as likely to have the reasons for requiring dose reduction of edoxaban, such as CrCl 30-50 ml/min (30.0% and 18.2%, respectively), weight ≤60 kg (30.6% and 7.8%, respectively), or concomitant use of verapamil or quinidine (P-gp inhibitors, 6.6% and 3.3%, respectively). This study is aimed to evaluate the safety of the low dose edoxaban therapy in patients with high bleeding risk and non-valvular AF in the real world population of Korea.

DETAILED DESCRIPTION:
The efficacy and safety of edoxaban has not been adequately studied in Asians versus non-Asians, who are quite different physiologically from each other. Although 1,943 patients from East Asia (1,010 were from Japan, 469 from China, 234 from Taiwan, and 230 from South Korea) were included in ENGAGE AF-TIMI 48, majority of the patient (19,162) were from non-East Asia. Compared with non-East Asian patients, the East Asia patients were twice as likely to have the reasons for requiring dose reduction of edoxaban, such as CrCl 30-50 ml/min (30.0% and 18.2%, respectively), weight ≤60 kg (30.6% and 7.8%, respectively), or concomitant use of verapamil or quinidine (P-gp inhibitors, 6.6% and 3.3%, respectively). Due to the relatively small number of patients in the East Asian group included in the analysis compared with that of the patients in the non-East Asian group, a limitation preventing it from providing sufficient power for such comparison is unavoidable. This study is aimed to evaluate the safety of the low dose edoxaban therapy in patients with high bleeding risk and non-valvular AF in the real world population of Korea.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation low dose edoxaban

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AF patients who are taking low dose edoxaban
Sampling Method: Non-Probability Sample
Enrollment: 2562 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
ISTH bleeding | through study completion, an average of 1 year
  ISTH bleeding

SECONDARY OUTCOMES:
non-major bleeding events | through study completion, an average of 1 year
  non-major bleeding events
Cardiovascular events | through study completion, an average of 1 year
  death, stroke, embolism, any bleeding
any side effect | through study completion, an average of 1 year
  any side effect

CONTACTS AND LOCATIONS:
Overall Officials: Young Keun On, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim JY, Kim J, Park SJ, Park KM, Han SJ, Kim DK, Park YM, Lee SH, Park JS, On YK; LEDIOS Registry Investigators. Optimal Dose of Edoxaban for Very Elderly Atrial Fibrillation Patients at High Risk of Bleeding: The LEDIOS Registry. Korean Circ J. 2024 Jul;54(7):398-406. doi: 10.4070/kcj.2024.0084. Epub 2024 May 10. PMID 38859644
- [Derived] Kim JY, Choi EK, Lim HE, Oh YS, Cho Y, On YK. Outcomes of On-Label Reduced-Dose Edoxaban in Patients With Atrial Fibrillation: The LEDIOS Registry. J Korean Med Sci. 2022 Dec 12;37(48):e335. doi: 10.3346/jkms.2022.37.e335. PMID 36513051